CLINICAL TRIAL: NCT01986621
Title: Identification of Patients at Higher Risk for Myocardial Injury or Type 4a Infarction Following Elective Coronary Artery Stenting
Brief Title: Myocardial Injury After Elective Coronary Stenting
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Haitham Abu Sharar, Physician, University Hospital Heidelberg
Other Study IDs: PCI MI4a
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Cardiac troponin; Antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing elective PCI

SUMMARY:
This pilot study aims to identify patients at moderate to high risk for peri-procedural (type 4) myocardial infarction or injury after after undergoing an elective coronary intervention (PCI) as measured by high sensitivity troponin T, who might benefit from more potent antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unknown coronary artery disease (CAD)
* Elective coronary intervention
* Minimum age of 18

Exclusion Criteria:

* Present acute coronary syndrome (ACS)
* Age under 18
* Pregnancy
* Any additional invasive intervention with potential myocardial injury
* Non ACS conditions responsible for elevation of cardiac troponin, such as acute pulmonary artery embolism, myocarditis or tachycardia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unknown CAD undergoing elective coronary intervention without receiving additional examination, such as biopsy, Ablation or any other procedure that could lead to myocardial injury resulting in elevation of the cardiac Troponin.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Postprocedural myocardial infarction (type 4a) or injury | up to 72 hours after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Abu Sharar, Dr. med., Principal Investigator — University Hospital Heidelberg; Evangelos Giannitsis, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Department of Cardiology - University Hospital of Heidelberg, Heidelberg, Germany